CLINICAL TRIAL: NCT01786720
Title: Analysis of the Time Taken for Newly Diagnosed COPD Patients to be Prescribed Triple Therapy
Brief Title: Analysis of the Time Taken to Triple Therapy (NOVARTIS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R04512
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: COPD
Keywords: COPD; Triple Therapy; ICS; LABA; LAMA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prior Triple Therapy: Patients prescribed triple therapy prior to initial date of COPD diagnosis
- Triple therapy at COPD diagnosis: Patients prescribed triple therapy on date of initial COPD diagnosis
- Triple therapy after COPD diagnosis: Patients prescribed triple therapy after initial date of COPD diagnosis

SUMMARY:
The proposed study will evaluate (for newly diagnosed Chronic Obstructive Pulmonary Disease (COPD) patients)the time taken to prescription of triple therapy by aiming to answer these following research questions:

1. The percentage of patients prescribed triple therapy, and when they first started receiving triple therapy.
2. For patients prescribed triple therapy, the time taken to triple therapy from initial diagnosis of COPD.
3. The variation in treatment pathways.
4. The factors associated with time taken to triple therapy.

DETAILED DESCRIPTION:
Triple therapy consists of long-acting beta agonist (LABA) + inhaled corticosteroids (ICS) + long-acting muscarinic antagonist (LAMA) and typically should be reserved for patients who have severe to very severe (FEV1 <50%) COPD symptoms or for patients who have two or more exacerbations per year. However previous research from RiRL indicate that 50% of patients at GOLD stage II (moderate) receive ICS of which half were on triple therapy.

To allow for multiple analysis regarding the factors that influence the likelihood of being prescribed triple therapy, a bespoke COPD dataset will be created to include:

1. Disease severity markers:
2. Confirmation of a COPD diagnosis at initial date of COPD diagnosis
3. Standard co-morbidities fields
4. Demographic fields

This retrospective, observational study using data of COPD patients will assess treatment pathways (changes/step up) from initial date of COPD diagnosis with the prescription of triple therapy as the endpoint.

Specific questions that will be asked are:

1. Does the percentage of COPD patients prescribed triple therapy vary dependent on time of initial date of COPD diagnosis?
2. Does the time taken to the prescription of triple therapy vary dependent on initial date of COPD diagnosis?

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥40 years at initial date of COPD diagnosis
* COPD diagnosis with Quality Outcome Framework (QoF) approved read code
* has spirometry data supportive of a COPD diagnosis in the 5 years around initial date diagnosis of COPD (FEV1 % predicted)
* Patient has one year of data prior to initial date of COPD diagnosis
* Patient has a minimum of two years of data post initial date of COPD diagnosi

Exclusion Criteria:

* Patients whose initial date of COPD diagnosis is before 1997

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have a QoF approved COPD read code and must be aged ≥ 40.
Sampling Method: Non-Probability Sample
Enrollment: 20154 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Triple Therapy Status | 1 year
  The proportion of patients prescribed triple therapy and whether they were prescribed it prior to, at, or after initial date of COPD diagnosis.
Initial date of COPD diagnosis | 1 year
  The date that patients were initially diagnosed with COPD. Categorised into cohorts- 1997-2001, 2002-2006, 2007-2010.

SECONDARY OUTCOMES:
Lung function grade | 1 year
  Patient lung function grade, calculated by GOLD I, II, III, IV criteria.
Asthma Diagnosis | 1 year
  Proportion of patients with a co-morbid asthma diagnosis
COPD patient group | 1 year
  Patients COPD patient group, calculated by GOLD A, B, C, D criteria dependent on symptoms and risk of patient.
COPD exacerbations (Clinical experience based) | 1 year
  Number of the following: (i) Asthma/copd-related*: a. Hospital attendance / admissions OR b. A&E attendance OR (ii) GP consultations for lower respiratory related tract infections
Smoking Status | 1 year
  Patient smoking status, taken from routine and questionnaire data
BMI | 1 year
  Patient BMI class
COPD co-morbidities | 1 year
  COPD co-morbidities are identified via Read codes that are recorded at any time.
  Co-morbidities are: GERD, Rhinitis, Heart Failure, Ischaemic Heart Disease, Diabetes, Osteoporosis, Chronic Renal Failure, Chronic Kidney Disease and Anxiety-Depression

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Research in Real Life Ltf, Cambridge, United Kingdom

REFERENCES:
- [Background] Price D, Yawn B, Brusselle G, Rossi A. Risk-to-benefit ratio of inhaled corticosteroids in patients with COPD. Prim Care Respir J. 2013 Mar;22(1):92-100. doi: 10.4104/pcrj.2012.00092. PMID 23135217
- [Background] Price D, Crockett A, Arne M, Garbe B, Jones RC, Kaplan A, Langhammer A, Williams S, Yawn BP. Spirometry in primary care case-identification, diagnosis and management of COPD. Prim Care Respir J. 2009 Sep;18(3):216-23. doi: 10.4104/pcrj.2009.00055. PMID 19688142